CLINICAL TRIAL: NCT02103439
Title: Multicenter Open-label Randomized, Comparative Clinical Study to Evaluate Efficacy and Safety of Algeron (Cepeginterferon Alfa-2b, CJSC "BIOCAD", Russia) With Ribavirin Compared to PegIntron (Peginterferon Alfa-2b, Schering-Plough Labo N.V., Belgium) With Ribavirin in Treatment of Chronic Hepatitis C in Human Immunodeficiency Virus-1 Infected Patients
Brief Title: An Open-label Randomized Multicenter Phase III Clinical Study Comparing Safety and Efficacy of Algeron (Cepeginterferon Alfa-2b) and and PegIntron (Peginterferon Alfa-2b) in Combination With Ribavirin as Combined Treatment of Chronic Hepatitis C in Human Immunodeficiency Virus-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-016-4
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis; Hepatitis C; Hepatitis C/ Human Immunodeficiency Virus Coinfection
Keywords: Hepatitis C; Cepeginterferon alfa; Peginterferon; Treatment
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Algeron (Experimental): Algeron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg)
  Interventions: Drug: Algeron
- PegIntron (Active Comparator): PegIntron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg).
  Interventions: Drug: PegIntron

INTERVENTIONS:
Drug: Algeron — 1.5 µg/kg of body weight subcutaneously, once a week
  Other Names: Cepeginterferon alfa-2b
  Arms: Algeron
Drug: PegIntron — 1.5 µg/kg of body weight subcutaneously, once a week
  Other Names: peginterferon alfa-2b
  Arms: PegIntron

SUMMARY:
The purpose of the study is to demonstrate the noninferiority of Algeron in combination with ribavirin compared to PegIntron in combination with ribavirin in treatment of chronic hepatitis C in Human Immunodeficiency Virus-1 infected patients

DETAILED DESCRIPTION:
The course of treatment in both groups shall be 12 weeks, and efficacy analysis, i.e. rate of rapid (after the 4th week) and early (after the 12th week) virologic response will be based on polymerase chain reaction data. For patients with treatment failure after the 12th week the antiviral therapy shall be discontinued. All patients who require further anti-viral treatment will receive a combination treatment with Algeron / PegIntron and ribavirin for another 36 weeks. Sustained virologic response will be assessed 24 weeks after last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Chronic hepatitis C (genotypes 1а, 1b, 2, 3, 4) confirmed by positive result of hepatitis C virus ribonucleic acid during > 6 months before screening visit or accompanied with increase in alanine aminotransferase (ALT) level > 6 months before screening visit.
* Confirmed Human Immunodeficiency Virus-1 infection based on enzyme-linked immunosorbent assay and immune blotting results.
* Clinically sustained phase of Human Immunodeficiency Virus-1 infection with absence of active opportunistic Human Immunodeficiency Virus-associated diseases for at least 30 calendar days before inclusion in the study.
* Level of CD4+-lymphocytes is not less than 500 cells/mm3 for patients not requiring highly active antiretroviral therapy and which will not be assigned to antiretroviral therapy during the study period.
* For patients receiving sustained highly active antiretroviral therapy for not less than 12 weeks and planning to continue comply with this treatment regimen during the following 24 weeks, level of CD4+-lymphocytes ≥300 cells/mm3, Human Immunodeficiency Virus ribonucleic acid ≤50 copies/ml.
* Men and women aged 18 to 70 inclusively.
* Body mass index in the range of 18 - 30 kg/m2 inclusively .
* Preserved protein-synthetizing liver function (International Normalized Ratio < 1.7, albumin > 35 g/l).
* Absence of signs of hepatic encephalopathy and ascites according to clinical examination and ultrasound examination.
* Patients with preserved child-bearing potential and their partners agree to use barrier method of contraception during the whole period of therapy and during 7 months after the treatment completion.
* Documentary confirmed results of liver elastography (fibroscan) during last year before enrollment in the study or patient agreement to undergo this examination during screening.

Exclusion Criteria:

* Intolerance of alfa-interferons, ribavirin or any components of tested drug product based on medical history.
* Presence of hepatitis B, A, E markers.
* Presence of documentary confirmed clinically significant concurrent liver diseases (alcoholic liver cirrhosis, drug-induced liver cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis, biliary cirrhosis etc.).
* Past history of Hepatitis C Virus treatment with interferon alfa or pegylated interferon alfa.
* For patients receiving sustained highly active antiretroviral therapy - presence of nevirapine, stavudine, zidovudine, didanosine in treatment regimen.
* Use of injectable and non-injectable interferons alfa/ interferon inducers for any indication (except for hepatitis C), radiotherapy, cytotoxic chemotherapy for one month prior to inclusion in the study.
* Cholestic hepatitis (level of direct bilirubin, alkaline phosphatase, gamma glutamyltransferase, exceeding upper normal limit in > 5 times).
* Decompensated liver cirrhosis confirmed with results of laboratory analyses (Child-Pugh class B, C) or ultrasound examination.
* Any documentary confirmed autoimmune diseases (such as Crohn's disease, ulcerative colitis, systemic lupus erythematosus, idiopathic thrombocytopenic purpura, scleroderma, autoimmune hemolytic anemia, severe psoriasis).
* Deviations of hematologic (hemoglobin less than lower normal limit; neutrophils < 1.5 x 10^9/l; thrombocytes < 90 x 10^9/ l) and biochemical (creatinine level > 1.5 times higher upper normal limit, ALT is > 10 times higher upper normal limit) parameters.
* Documentary confirmed diagnosis of hemoglobinopathy (for example, thalassemia, sickle-cell anemia).
* Severe depression, schizophrenia, any other mental disorders which according to the investigator are contraindications for antiviral treatment.
* Epilepsy and/or central nervous system disorder.
* Disorder of thyroid function (level of thyroid stimulating hormone out of the normal range).
* Documentary confirmed or suspected hepatocellular carcinoma based on the results of alfa-fetoprotein (AFP) assay ≥ upper normal limit.
* Antinuclear antibodies (ANA) titer measured at screening is not less than 1:640 or documentary confirmed signs of autoimmune hepatitis based on the results of biopsy.
* Documentary confirmed malignant neoplasms.
* Documentary confirmed lung diseases associated with respiratory failure.
* Treatment of Human Immunodeficiency Virus-1 with immunotherapeutic vaccines within 90 days prior to screening.
* Necessity in assignment of antimycobacterial therapy.
* Pregnancy, lactation period.
* Documentary confirmed retinopathy (for example, cytomegalovirus retinitis, macular degeneration).
* Severe concurrent diseases (for example, severe arterial hypertension, sever coronary heart disease, heart failure, decompensated diabetes mellitus and other) which are contraindications for antiviral therapy according to the investigator opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2015-08-26 (Actual); Study Completion 2015-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Moshkovich, M.D., Principal Investigator — State Institution of Nizhny Novgorod region "Regional Center for Prevention and Control of AIDS and other infectious diseases"; Firaya Nagimova, PhD, Principal Investigator — State Public Healthcare Institution National Center for the Prevention and Control of AIDS and other infectious diseases of the Ministry of Health of the Republic of Tatarstan; Oleg Kozyrev, PhD, Principal Investigator — State Healthcare Institution "Volgograd Regional Center for the Prevention and Control of AIDS and infectious diseases"; Andrey Shuldyakov, M.D., PhD, Principal Investigator — State Budgetary Higher Vocational Education Institution V.I. Razumovsky Saratov State University of medicine; Vadim Rassokhin, PhD, Principal Investigator — State Healthcare Institution Center for the Prevention and Control of AIDS and infectious diseases of the city, St.Petersburg CityHealth Department; Lidia Sklar, M.D., PhD, Principal Investigator — State Budgetary Higher Vocational Education Institution Pacific State Medical University, Ministry of Health of the Russian Federation
Locations (6):
- Russia (6):
  - State Public Healthcare Institution National Center for the Prevention and Control of AIDS and other infectious diseases of the Ministry of Health of the Republic of Tatarstan, Kazan', Tatarstan Republic
  - State Institution of Nizhny Novgorod region "Regional Center for Prevention and Control of AIDS and other infectious diseases", Nizhny Novgorod
  - State Healthcare Institution Center for the Prevention and Control of AIDS and infectious diseases of the city, St.Petersburg CityHealth Department, Saint Petersburg
  - State Budgetary Higher Vocational Education Institution V.I. Razumovsky Saratov State University of medicine, Saratov
  - State Budgetary Higher Vocational Education Institution Pacific State Medical University, Ministry of Health of the Russian Federation, Vladivostok
  - State Healthcare Institution "Volgograd Regional Center for the Prevention and Control of AIDS and infectious diseases", Volgograd

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Algeron | PegIntron
Started | 70 | 70
Completed | 67 | 67
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Algeron | PegIntron | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [30 to 37] | 34 [31 to 37] | 33.5 [31 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 45 | 46 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 68 | 69 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Early Virological Response
Description: Proportion of randomized patients achieving early virologic response - negative polymerase chain reaction result for Hepatitis C Virus ribonucleic acid (< 15 IU/ml) or ≥ 2log10 decrease of viral load after 12 weeks of study treatment
Time Frame: 12 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Algeron | PegIntron
Number analyzed (Participants) | 70 | 70
percentage of patients | 90.0 | 81.4
Statistical Analysis 1: Comparison: Algeron vs PegIntron; Test type: Non-Inferiority or Equivalence — the lower limit of the 95% confidence interval for the difference in proportions between the difference in the early virological response rate with Algeron and PegIntron should be higher than the non-inferiority margin of 0.2 (-20%); p = 0.227, Fisher Exact

2. Secondary Outcome: Rapid Virological Response
Description: Proportion of randomized patients achieving rapid virologic response - negative polymerase chain reaction result for Hepatitis C Virus ribonucleic acid (< 15 IU/ml) after 4 weeks of treatment
Time Frame: 4 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Algeron | PegIntron
Number analyzed (Participants) | 70 | 70
percentage of patients | 51.4 | 37.1
Statistical Analysis 1: Comparison: Algeron vs PegIntron; Test type: Non-Inferiority or Equivalence — the lower limit of the 95 % confidence interval between the difference in rate of rapid virological response with Algeron and PegIntron should be more than the non-inferiority margin (-20 %); p > 0.05, Fisher Exact

3. Secondary Outcome: Rapid Virological Response in Patients With Different Hepatitis C Virus Genotypes
Description: Proportion of randomized patients with different Hepatitis C Virus (HCV) genotypes achieving rapid virological response - negative polymerase chain reaction result for HCV ribonucleic acid (< 15 IU/ml) after 4 weeks of treatment
Time Frame: 4 weeks
Measure: Number; unit: percentage of patients
Groups:
- Algeron - HCV-1: Patients with HCV genotype 1, received Algeron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg)
  Algeron: 1.5 µg/kg of body weight subcutaneously, once a week
- Algeron - HCV-2/3: Patients with HCV genotype 2 or 3, received Algeron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg)
  Algeron: 1.5 µg/kg of body weight subcutaneously, once a week
- PegIntron - HCV-1: Patients with HCV genotype 1, received PegIntron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg).
  PegIntron: 1.5 µg/kg of body weight subcutaneously, once a week
- PegIntron - HCV-2/3: Patients with HCV genotype 2 or 3, received PegIntron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg).
  PegIntron: 1.5 µg/kg of body weight subcutaneously, once a week
Arm/Group | Algeron - HCV-1 | Algeron - HCV-2/3 | PegIntron - HCV-1 | PegIntron - HCV-2/3
Number analyzed (Participants) | 34 | 36 | 33 | 37
percentage of patients | 23.5 | 77.8 | 21.2 | 51.4

4. Secondary Outcome: Viral Breakthrough
Description: Proportion of patients in each groups with level of Hepatitis C Virus ribonucleic acid > 15 IU/ml after Hepatitis C Virus ribonucleic acid was not present or Hepatitis C Virus ribonucleic acid was increased by more than 1log10 from baseline at 4 or 12 weeks of treatment
Time Frame: screening data and at 4 or 12 weeks of treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Algeron | PegIntron
Number analyzed (Participants) | 70 | 70
percentage of patients | 0 | 0

5. Primary Outcome: Early Virological Response in Patients With Different Hepatitis C Virus Genotypes
Description: Proportion of randomized patients with different Hepatitis C Virus (HCV) genotypes achieving early virologic response - negative polymerase chain reaction result for HCV ribonucleic acid (< 15 IU/ml) or ≥ 2log10 decrease of viral load after 12 weeks of study treatment
Time Frame: 12 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Algeron - HCV-1 | Algeron - HCV-2/3 | PegIntron - HCV-1 | PegIntron - HCV-2/3
Number analyzed (Participants) | 34 | 36 | 33 | 37
percentage of patients | 82.4 | 97.2 | 75.8 | 88.5

6. Secondary Outcome: Biochemical Response
Description: Proportion of patients in each group with alanine aminotransferase level ≤ upper normal limit after 12 weeks of therapy
Time Frame: 12 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Algeron | PegIntron
Number analyzed (Participants) | 70 | 70
percentage of patients | 68.6 | 82.9

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The number of patients for the efficacy analysis was 140 patients. 141 patients were included in the safety analysis, including 1 patient in PegIntron group withdrawn at early stages due to a violation of inclusion/non-inclusion criteria [previous AVT cycle], who was not considered to be enrolled in the study due to serious protocol violation.
Groups:
- PegIntron: PegIntron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg).
  PegIntron: 1.5 µg/kg of body weight subcutaneously, once a week
  The safety analysis included 71 patients received at least 1 dose of PegIntron (taking into account one patient withdrawn at early stages of the study due to a protocol violation [previous treatment of hepatitis C with interferon alfa], who was withdrawn from the mITT-analysis)
Arm/Group | Algeron | PegIntron
Serious Adverse Events (participants affected / at risk) | 0/70 | 2/71
Other Adverse Events (participants affected / at risk) | 70/70 | 69/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Algeron (N=70) | PegIntron (N=71)
CTCAE 4.03 Grade 4 anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
cavitary pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Algeron (N=70) | PegIntron (N=71)
Flu-like syndrome (General disorders) | 38 (46) | 41 (87)
Asthenia (weakness, fatigue) (General disorders) | 17 (25) | 16 (23)
Headache (Nervous system disorders) | 12 (38) | 13 (25)
Irritability, emotional lability (Psychiatric disorders) | 4 (4) | 4 (4)
Sleep disorders (Nervous system disorders) | 4 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (21) | 2 (8)
Stomach pain (Gastrointestinal disorders) | 7 (9) | 5 (5)
Decreased appetite (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 6 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (16) | 3 (6)
Skin itch (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2)
Skin redness (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Skin dryness and exfoliation (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Leucopenia (Blood and lymphatic system disorders) | 60 (67) | 59 (69)
Neutropenia (Blood and lymphatic system disorders) | 53 (67) | 51 (66)
Lymphopenia (Blood and lymphatic system disorders) | 43 (52) | 55 (62)
Decreased level of CD4+ lymphocytes (Blood and lymphatic system disorders) | 8 (8) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 39 (39) | 36 (37)
Need in filgrastim (Blood and lymphatic system disorders) | 8 (8) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 49 (50) | 57 (59)
Need in Rebetol dose correction due to anemia (Blood and lymphatic system disorders) | 12 (12) | 11 (11)
Hyperbilirubinaemia (Hepatobiliary disorders) | 22 (27) | 26 (28)
Direct bilirubin increased (Hepatobiliary disorders) | 31 (33) | 31 (34)
Increased albumin (Hepatobiliary disorders) | 16 (17) | 25 (29)
Increased alanine aminotranferase (Hepatobiliary disorders) | 25 (26) | 18 (18)
Increased aspartate aminotranferase (Hepatobiliary disorders) | 28 (32) | 29 (31)
Increased gamma glumamyltransferase (Hepatobiliary disorders) | 21 (21) | 31 (36)
Increased alkaline phosphotase (Hepatobiliary disorders) | 7 (7) | 6 (6)
Hyperglycemia (Endocrine disorders) | 6 (6) | 8 (8)
Hypoglycemia (Endocrine disorders) | 10 (12) | 14 (15)
Increased triglycerides (Metabolism and nutrition disorders) | 34 (38) | 37 (42)
Increased cholesterol (Metabolism and nutrition disorders) | 11 (12) | 17 (17)
Increased thyroid stimulating hormone (Endocrine disorders) | 4 (4) | 2 (2)
Increased creatinine (Renal and urinary disorders) | 11 (11) | 6 (6)
Hyperemia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No